CLINICAL TRIAL: NCT04524962
Title: Phase I/IIA Study of Descartes-30 in Acute Respiratory Distress Syndrome
Brief Title: Study of Descartes-30 in Acute Respiratory Distress Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 1 enrollment completed. Further clinical development terminated
Sponsor: Cartesian Therapeutics (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC30-1A; 5R44HL158446 (NIH); 2021-MSCRFCL-5 (Other Grant/Funding Number: Maryland Stem Cell Research Foundation)
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Acute Respiratory Distress Syndrome; Covid19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Descartes 30 (Experimental)
  Interventions: Biological: Descartes 30

INTERVENTIONS:
Biological: Descartes 30 — Mesenchymal Stem Cells or MSCs RNA-engineered to secrete a combination of DNases.

SUMMARY:
Emergency study to test the safety of Descartes-30 cells in patients with moderate-to-severe acute respiratory distress syndrome (ARDS) AND COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older at the time of enrollment
* Patient maintains a diagnosis of moderate or severe ARDS according to the Berlin definition of ARDS

Exclusion Criteria:

* Patient is currently enrolled into another therapeutic clinical trial with an experimental therapy that has not received marketing approval by U.S. FDA.
* Patient is in moribund state with expected survival <24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Medical Center Medical Center, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Descartes 30: Dose Level 1: Participants were administered 100 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
- Descartes-30: Dose Level 2: Participants were administered 300 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
- Descartes-30: Dose Level 3: Participants were administered 600 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
- Descartes-30: Dose Level 4 Cells/Infusion: Participants were administered 1200 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
Period: Overall Study
Arm/Group | Descartes 30: Dose Level 1 | Descartes-30: Dose Level 2 | Descartes-30: Dose Level 3 | Descartes-30: Dose Level 4 Cells/Infusion
Started | 3 | 3 | 5 | 1
Completed | 3 | 3 | 5 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Descartes 30 Dose Level 1: Participants were administered 100 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
- Descartes 30 Dose Level 2: Participants were administered 300 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
- Descartes 30 Dose Level 3: Participants were administered 600 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
- Descartes 30 Dose Level 4: Participants were administered 1200 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
- Total: Total of all reporting groups
Arm/Group | Descartes 30 Dose Level 1 | Descartes 30 Dose Level 2 | Descartes 30 Dose Level 3 | Descartes 30 Dose Level 4 | Total
Number analyzed (Participants) | 3 | 3 | 5 | 1 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 0 | 8
  >=65 years | 0 | 1 | 2 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 4
  Male | 1 | 2 | 4 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 2 | 4 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 3 | 1 | 5 | 1 | 10
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 3 | 5 | 1 | 10
  Turkey | 2 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Safety of Descartes-30 in Patients With Moderate-to-severe ARDS.
Description: Safety will be determined principally by assessment of adverse events (AEs) and serious adverse events (SAEs).
Time Frame: 3 months
Measure: Number; unit: treatment related adverse events
Groups:
- Descartes-30: Dose Level 4: Participants were administered 1200 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
Arm/Group | Descartes 30: Dose Level 1 | Descartes-30: Dose Level 2 | Descartes-30: Dose Level 3 | Descartes-30: Dose Level 4
Number analyzed (Participants) | 3 | 3 | 5 | 1
treatment related adverse events | 1 | 1 | 3 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, up to 3 months.
Groups:
- Descartes 30: Dose Level 2: Participants were administered 300 million cells of Descartes-30 via intravenous catheter on Days 0, 1, 2.
Arm/Group | Descartes 30: Dose Level 1 | Descartes 30: Dose Level 2 | Descartes-30: Dose Level 3 | Descartes-30: Dose Level 4
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 2/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 3/5 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 5/5 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Descartes 30: Dose Level 1 (N=3) | Descartes 30: Dose Level 2 (N=3) | Descartes-30: Dose Level 3 (N=5) | Descartes-30: Dose Level 4 (N=1)
Sepsis (Immune system disorders) | 1 | 0 | 0 | 0 — Not related to Descartes-30
Intubation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Not related to Descartes-30
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 0 — Not related to Descartes-30
Cardiopulmonary arrest (Cardiac disorders) | 0 | 0 | 1 | 0 — Not related to Descartes-30
Acute kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 — Not related to Descartes-30
Acute leg ischemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — Not related to Descartes-30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Descartes 30: Dose Level 1 (N=3) | Descartes 30: Dose Level 2 (N=3) | Descartes-30: Dose Level 3 (N=5) | Descartes-30: Dose Level 4 (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 — Possibly related to Descartes-30
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 | 1 (2) | 0 — Possibly related to Descartes-30
Fever (Immune system disorders) | 1 (1) | 1 (1) | 0 | NA — Possibly related to Descartes-30
Blood stream infection (Blood and lymphatic system disorders) | 1 (2) | 0 | 0 | 0 — Not related to Descartes-30
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 — Not related to Descartes-30
Sepsis (Infections and infestations) | 1 | 1 | 2 | NA — Not related to Descartes-30
Mucosal bleeding (Infections and infestations) | 1 | 0 | 0 | 0 — Not related to Descartes-30
MRSA pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Not related to Descartes-30
UTI (Renal and urinary disorders) | 1 | 0 | 0 | 0 — Not related to Descartes-30
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Not related to Descartes-30
Steroid Induced hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Not related to Descartes-30
ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 — Not related to Descartes-30
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Not related to Descartes-30
Creatinine increased (Investigations) | 0 | 1 | 3 | NA — Not related to Descartes-30
INR increased (Investigations) | 0 | 0 | 1 | 0 — Not related to Descartes-30
AST increased (Investigations) | 0 | 0 | 1 | 0 — Not related to Descartes-30
ALT increased (Investigations) | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — Not related to Descartes-30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04524962/Prot_SAP_000.pdf